CLINICAL TRIAL: NCT06737042
Title: EFFICACY and SAFETY of GZR18 INJECTED EVERY 2 WEEKS (Q2W) in PARTICIPANTS WITHOUT TYPE 2 DIABETES, WHO HAVE OBESITY or ARE OVERWEIGHT: a RANDOMIZED, TIRZEPATIDE- and PLACEBO-CONTROLLED STUDY
Brief Title: Efficacy and Safety of GZR18 Every 2 Weeks Versus Tirzepatide and Placebo in Obese or Overweight Participants
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GL-GLP-2001
Record Dates: First submitted 2024-12-16; First posted 2024-12-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: GLP-1, Obesity, Overweight, Weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 24 mg GZR18 group (Experimental): 24 mg GZR18 group: 76 participants (57 receiving GZR18 and 19 receiving placebo)
  Interventions: Drug: GZR18
- 36 mg GZR18 group (Experimental): 36 mg GZR18 group: 76 participants (57 receiving GZR18 and 19 receiving placebo)
  Interventions: Drug: GZR18
- 48 mg GZR18 group (Experimental): 48 mg GZR18 group: 76 participants (57 receiving GZR18 and 19 receiving placebo)
  Interventions: Drug: GZR18
- Tirzepatide group (Active Comparator): Tirzepatide group: 57 participants receiving 15 mg tirzepatide
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: GZR18 — GLP-1
  Arms: 24 mg GZR18 group; 36 mg GZR18 group; 48 mg GZR18 group
Drug: Tirzepatide — Active Comparator
  Arms: Tirzepatide group

SUMMARY:
This is a Phase 2 study to evaluate the safety and efficacy of 24, 36, and 48 mg GZR18 (Q2W) compared with placebo and 15 mg tirzepatide (QW). The study will evaluate weight management in participants with obesity (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with weight-related comorbidities (excluding type 2 diabetes mellitus).

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, randomized, parallel-group, partially-blinded, placebo and tirzepatide-controlled study of the safety and efficacy of 24, 36, and 48 mg GZR18 (Q2W) compared with placebo and 15 mg tirzepatide (QW). The study will evaluate weight management in participants with obesity (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with weight-related comorbidities (excluding type 2 diabetes mellitus).

The study will comprise a 2-week screening period (Days -14 to -1), a 36-week treatment period (Weeks 0 to 36), which includes a titration period and a maintenance dose period, and a safety follow-up period of 2 weeks after the primary endpoint assessment (ie, 4 weeks after the last GZR18 dose and 3 weeks after the last tirzepatide dose).

Approximately 285 participants will be randomized at Week 0 into 1 of 4 groups, stratified by sex. The study will be partially-blinded (intragroup blinded); treatment in the GZR18 groups will be blinded (GZR18 vs placebo), but GZR18 vs tirzepatide will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age (both inclusive) at the time of signing the informed consent form (ICF).
2. History of failing to lose sufficient weight with lifestyle/dietary modification.

BMI ≥30.0 kg/m2, or

BMI ≥27.0 kg/m2 with at least 1 of the following:

* Hypertension: defined as taking blood pressure (BP) lowering medication or have a systolic blood pressure (SBP) of ≥130 mmHg or a diastolic blood pressure (DBP) of ≥80 mmHg at screening.
* Dyslipidemia: defined as taking lipid-lowering medication or have LDL ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein (HDL) <40 mg/dL (1.0 mmol/L) for men or HDL <50 mg/dL (1.3 mmol/L) for women at screening.
* Obstructive sleep apnea.
* Cardiovascular disease: defined as having eg, ischemic cardiovascular disease or New York Heart Association (NYHA) Functional Classification Class I to II heart failure.

  4. In the investigator's opinion, are well motivated, capable, and willing to:
* Learn how to self-inject the IP as required for this protocol (visually impaired persons who are not able to perform the injections must have the assistance of a sighted individual trained to inject the IP; persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject the IP).
* Inject the IP (or receive an injection from a trained individual if visually impaired or with physical limitations).
* Follow study procedures for the duration of the study, including, but not limited to, lifestyle advice (eg, dietary changes and physical activity plan), complete the electronic diary (eDiary), and complete required questionnaires.
* Identify the biological sex for the study stratification. 5.Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Medical Conditions Related to Obesity

1. A self-reported change (increase or decrease) in body weight >5 kg within 3 months prior to screening.
2. Prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to screening).
3. Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 6 months prior to screening, including but not limited to:

   * Mucosal ablation
   * Gastric artery embolization
   * Intragastric balloon
   * Duodenal-jejunal endoluminal liner Related to Diabetes
4. History of type 1 or T2DM, history of ketoacidosis, or hyperosmolar state/coma.
5. At least 1 laboratory value suggestive of diabetes during screening, including 1 or more of HbA1c ≥6.5% (48 mmol/mol), fasting serum glucose ≥126 mg/dL (7.0 mmol/L), or random glucose ≥200 mg/dL (11.1 mmol/L).

   Other Medical Conditions
6. Renal impairment measured as estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2, calculated by chronic kidney disease-epidemiology collaboration (CKD-EPI) as determined by central laboratory during screening.
7. Known clinically significant gastric emptying abnormality (eg, severe gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect GI motility.
8. History of acute or chronic pancreatitis. A participant with a history of acute pancreatitis caused by gallstones may be included in the study if the participant has a cholecystectomy to resolve the problem.
9. Thyroid-stimulating hormone (TSH) outside of the range of 0.4 to 6.0 mIU/L at screening.

   Note: Participants receiving treatment for hypothyroidism may be included, provided their thyroid hormone replacement dose has been stable for at least 6 months.

   Note: TSH values above the normal range can, in some participant, suggest subclinical hypothyroidism. If, in the investigator's opinion, the participant has subclinical hypothyroidism and may require initiation of thyroid hormone replacement during the study, the participant should be excluded from the study.
10. Obesity induced by other endocrinologic disorders (eg, Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (eg, melanocortin 4 receptor deficiency or Prader-Willi syndrome).
11. History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder (eg, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 years.

    Note: Participants with MDD or generalized anxiety disorder whose disease state is considered stable for the past 2 years and expected to remain stable throughout the course of the study, in the opinion of the investigator, may be considered for inclusion if they are not on excluded medications.
12. A history of suicide attempt.
13. Patient health questionnaire-9 (PHQ-9) score of 15 or more at screening.
14. On the Columbia Suicide Severity Rating Scale (C-SSRS) prior to randomization:

    * a "yes" answer to Question 4 (active suicidal ideation with some intent to act, without specific plan) on the "suicidal ideation" portion of the C-SSRS or
    * a "yes" answer to Question 5 (active suicidal ideation with specific plan and intent) on the "suicidal ideation" portion of the C-SSRS or
    * a "yes" answer to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act, or behavior) on the "suicidal behavior" portion of the C-SSRS and
    * the ideation or behavior occurred within the past month
15. Uncontrolled hypertension (SBP ≥160 mmHg and/or DBP ≥100 mmHg). If a participant is on antihypertensive therapies, doses must be stable for 30 days prior to screening. For participants with uncontrolled hypertension at screening, antihypertensive medication may be started or adjusted. BP must meet the protocol criterion for hypertension control with stable treatment for at least 30 days before re-screening.
16. An elevated resting pulse rate >100 bpm at baseline.
17. Any of the following cardiovascular conditions within 3 months prior to screening:

    * Acute myocardial infarction
    * Cerebrovascular accident (stroke)
    * Unstable angina
    * Hospitalization due to congestive heart failure (CHF)
18. Ongoing or history of frequent intermittent or chronic tachyarrhythmia syndromes (eg, atrial fibrillation, supraventricular tachycardia, and positional orthostatic tachycardia syndrome).

    Note: Participants with a history of premature atrial contractions or premature ventricular contractions may be included.
19. NYHA Functional Classification III or IV CHF.
20. An electrocardiogram (ECG) considered by the investigator indicative of active cardiac disease or with abnormalities that may interfere with the interpretation of changes in ECG intervals at screening.
21. Acute or chronic hepatitis, or signs and symptoms of any other liver disease other liver disease except nonalcoholic fatty liver disease (NAFLD) (ie, participants with NAFLD are eligible for participation), or any of the following at screening:

    * alanine aminotransferase (ALT) >3 × the upper limit of normal (ULN)
    * alkaline phosphatase (ALP) >1.5 × ULN
    * total bilirubin level >1.5 × ULN (except for cases of known Gilbert's Syndrome)
22. Serum calcitonin level of:

    * 20 ng/L, if eGFR ≥60 mL/min/1.73 m2
    * 35 ng/L, if eGFR ≤60 mL/min/1.73 m2
23. A family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
24. A history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for <5 years.
25. Any other condition not listed in this section (eg, hypersensitivity or intolerance) that is a contraindication to GLP-1R agonists.
26. A history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the investigator, may preclude the participant from following and completing the protocol.
27. Alcohol consumption >14 units/week for women and >21 units/week for men.
28. A history of use of marijuana or tetrahydrocannabinol (THC)-containing products within 3 months of enrollment or unwillingness to abstain from marijuana or THC-containing product use during the study.

    Note: If a participant has used cannabidiol oil during the past 3 months but agrees to refrain from use for the duration of the study, the participant may be enrolled.
29. Have had an organ transplant (corneal transplants [keratoplasty] are allowed) or are awaiting an organ transplant.
30. Any hematological condition that may interfere with HbA1c measurements (eg,
31. A blood donation of ≥500 mL within the previous 8 weeks of screening or a blood transfusion or severe blood loss within the prior 3 months, or have known hemoglobinopathy, hemolytic anemia, sickle cell anemia, or a hemoglobin value <11 g/dL (men) or <10 g/dL (women), or any other condition known to interfere with HbA1c methodology.
32. A history of atopy (severe or multiple allergic manifestations) or clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, anaphylaxis, angioedema, or exfoliative dermatitis).
33. A fasting serum triglyceride level of >500 mg/dL at screening. If a participant is on lipid-lowering therapies, doses must be stable for 30 days prior to screening.

    Prior/Concomitant Therapy
34. Are receiving or have received within 3 months prior to screening chronic (>2 weeks) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, single intraarticular injection, or inhaled preparations) or have evidence of a significant, active autoimmune abnormality (eg, lupus or rheumatoid arthritis) that has required (within the last 3 months) or is likely to require, in the opinion of the investigator, concurrent treatment with systemic glucocorticoids (excluding topical, intraocular, intranasal, intraarticular, or inhaled preparations) during the course of the study.
35. Receiving treatment with or have a history of treatment with (within 3 months prior to screening) medications that may cause significant weight gain including, but not limited to, tricyclic antidepressants, atypical antipsychotics, and mood stabilizers:

    Examples:
    * imipramine
    * amitriptyline
    * mirtazapine
    * paroxetine
    * phenelzine
    * chlorpromazine
    * thioridazine
    * clozapine
    * olanzapine valproic acid and its derivatives
    * lithium Note: Selective serotonin reuptake inhibitors other than paroxetine are permitted.
36. Have taken within 3 months prior to screening medications (prescribed or over thecounter) or alternative remedies intended to promote weight loss.

    Examples include, but are not limited to:
    * Saxenda® (liraglutide 3.0 mg) or other GLP-1R agonists
    * Xenical®/Alli® (orlistat)
    * Meridia® (sibutramine)
    * Acutrim® (phenylpropanolamine)
    * Sanorex® (mazindol)
    * Adipex® or LomairaTM (phentermine)
    * QsymiaTM (phentermine/topiramate combination)
    * Contrave® (naltrexone/bupropion)
37. Use of metformin or any other glucose-lowering medication, whether prescribed for polycystic ovarian syndrome or diabetes prevention is not permitted.
38. Have started implantable or injectable contraceptives (such as Depo Provera®) within 18 months prior to screening.

    Prior/Concurrent Clinical Study Experience
39. Have known allergies to GLP-1R agonists or GZR18.
40. Are currently enrolled in any other clinical study involving an IP or any other type of medical research judged not to be scientifically or medically compatible with this study.
41. Within the last 30 days, participated in a clinical study and received treatment, whether active or placebo. If the study involved an IP, 5 half-lives or 30 days, whichever is longer, should have passed.
42. Have previously completed or withdrawn from this study or any other study investigating GZR18 and have previously received GZR18.

    Other Exclusions
43. Women of childbearing potential (WOCBP) who:

    * Are pregnant or intend to become pregnant (or have a positive pregnancy test at screening).
    * Are lactating/breastfeeding (including the use of a breast pump).
    * Are unwilling to remain abstinent or use acceptable birth control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 36 weeks
  To demonstrate that GZR18 24 mg, 36 mg, and 48 mg is superior to placebo based on percentage change in body weight after 36 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - KUR Research - Trinity @ Bessemer, AL Site Network, Bessemer, Alabama
  - KUR Research - Trinity @ Centreville Site Network, Centreville, Alabama
  - ERG - Woodland Int'l Research Group, Little Rock, Arkansas
  - ERG - Woodland Research Northwest, Rogers, Arkansas
  - Ark Clinical Research Ark-Fountain Valley, Fountain Valley, California
  - Ark Clinical Research Ark-Long Beach, Long Beach, California
  - Clinedge - Central Valley Research, LLC, Modesto, California
  - Populace Health, LLC - Catalina Research Institute, Montclair, California
  - East Coast Institute for Research - ECIR Jacksonville (Southside), Jacksonville, Florida
  - East Coast Institute for Research ECIR Jacksonville (Headquarters) University, Jacksonville, Florida
  - 3Sync Research - PCRS Network, Lake Worth, Florida
  - Clever Medical Research - PCRS Network, Miami, Florida
  - KUR Research @ Columbia Site Network, Columbia, Maryland
  - Populace Health, LLC - Elixia SISU, Springfield, Massachusetts
  - Populace Health, LLC - Vector Clinical Trials, Las Vegas, Nevada
  - Populace Health, LLC - CTI Clinical Research Center, Cincinnati, Ohio
  - ERG - Ohio Clinical Trials, Columbus, Ohio
  - Elligo Clinical Research Center - Austin, Austin, Texas
  - Clinvax Katy Research Center, Katy, Texas
  - Endeavor Clinical Trials, San Antonio, Texas